CLINICAL TRIAL: NCT01978587
Title: A Phase 1, Open-label, Sequential Crossover Study to Evaluate the Effect of Hemodialysis on the Pharmacokinetics of JTZ-951 in Subjects With End-stage Renal Disease
Brief Title: Effect of Hemodialysis on the PK of JTZ-951 in Subjects With End-stage Renal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AZ951-U-13-005
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Anemia in Chronic Kidney Disease
Keywords: End-stage Renal Disease; Hemodialysis; Pharmacokinetics
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — enarodustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose 1 JTZ-951 (Experimental): Tablets, 1 dose on Day 1 before hemodialysis
  Interventions: Drug: JTZ-951
- Dose 2 JTZ-951 (Experimental): Tablets, 1 dose on Day 8 after hemodialysis
  Interventions: Drug: JTZ-951

INTERVENTIONS:
Drug: JTZ-951

SUMMARY:
The purpose of this study is to evaluate the effect of hemodialysis on the pharmacokinetics (PK) of JTZ-951 and to evaluate the safety of 2 doses of JTZ-951 in subjects with end-stage renal disease (ESRD) receiving hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have ESRD and have been receiving maintenance hemodialysis for at least 12 weeks prior to the Screening Visit
* Body weight (post-dialysis weight) greater than 45.0 kg and a body mass index between 20.0 and 40.0 kg/m2 (inclusive) at the Screening Visit

Exclusion Criteria:

* Acute coronary syndrome (e.g., myocardial infarction) within 1 year prior to admission
* Uncontrolled hypertension at the Screening Visit or Day -1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum concentration) of JTZ-951 when administered before and after hemodialysis | Days 1 to 4 and 8 to 11
tmax (time to reach maximum concentration) of JTZ-951 when administered before and after hemodialysis | Days 1 to 4 and 8 to 11
AUC (area under the concentration-time curve) of JTZ-951 when administered before and after hemodialysis | Days 1 to 4 and 8 to 11
t1/2 (elimination half-life) of JTZ-951 when administered before and after hemodialysis | Days 1 to 4 and 8 to 11

SECONDARY OUTCOMES:
Number of subjects with adverse events | 14 days
Vital signs and ECG (electrocardiogram) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Hideyuki Yamamoto, Study Chair — Akros Pharma Inc.
Locations (1):
- Minneapolis, Minnesota, United States